CLINICAL TRIAL: NCT06654791
Title: A Phase I Clinical Study to Evaluate the Mass Balance of [14C]SIM0270 in Healthy Chinese Adult Subjects
Brief Title: Mass Balance Clinical Trial of SIM0270
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Collaborators: Nanjing Zaiming Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIM0270-103
Record Dates: First submitted 2024-10-21; First posted 2024-10-23 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Healthy Participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- [14C]SIM0270 group (Other): Single arm study
  Interventions: Drug: [14C] SIM0270 Oral Preparation

INTERVENTIONS:
Drug: [14C] SIM0270 Oral Preparation — Use according to the prescribed protocol

SUMMARY:
This is a single-center, non-randomized, open-label, single-cohort, single-dose phase I clinical study in healthy Chinese adult male subjects.

DETAILED DESCRIPTION:
The main objectives of this study were as follows:

1. To quantitatively analyze the total radioactivity in excreta of healthy subjects after a single oral administration of [14C]SIM0270, and to obtain the data of human radioactive excretion rate and main excretion routes.
2. After a single oral administration of [14C]SIM0270 in healthy subjects, radioactive metabolite profiles in plasma, urine and feces were investigated to identify metabolites, and the metabolic pathway, main metabolites and elimination pathway of SIM0270 in human body were determined.
3. The total radioactivity in whole blood and plasma of healthy subjects after a single oral administration of [14C]SIM0270 was quantitatively analyzed, the pharmacokinetic characteristics of total radioactivity in plasma were evaluated, and the distribution of total radioactivity in whole blood and plasma was investigated.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects fully understand the test content, process and possible adverse reactions, voluntarily sign informed consent, have good communication with the researchers, and can complete all the test procedures in accordance with the protocol.
2. Chinese male, aged between 18 and 45 years old (including the critical value, subject to the signing of the informed consent).
3. Weight ≥50.0kg, and body mass index (BMI) between 19.0 and 26.0 kg/m2 (including the cut-off value).

Exclusion Criteria:

Clinical examination:

1. Patients who have undergone physical examination, vital signs, laboratory examination (blood routine, blood biochemistry, thyroid function, coagulation function, urine routine, stool analysis), vision and eye examination (slit-lamp, intraocular pressure and fundus photography), X-ray chest film (anterior and lateral), abdominal B-ultrasound (liver, bile, pancreas, spleen and kidney) and other abnormal examinations with clinical significance;
2. Patients with abnormal 12-lead ECG and clinical significance (including but not limited to: complete left bundle branch block; Right bundle branch block; First, second, or third degree heart block), or QTcF > 450 ms after correction using the Fridericia formula (QTcF=QT / {(60/ heart rate)^0.33});
3. Hepatitis B surface antigen, hepatitis C antibody, HIV antibody or syphilis antibody positive;

   Medication history:
4. Those who have used prescription drugs, non-prescription drugs, health drugs or live attenuated vaccines including western medicines or proprietary Chinese medicines within 14 days before the screening period;
5. Those who participated in any clinical trial and received the experimental drug or medical device intervention within 3 months prior to the screening period;
6. Any drug with a strong/medium acting inhibitor or a strong/medium acting inducer of CYP3A4 in the 4 weeks prior to enrollment (see Appendix 1).

   Disease history and surgical history:
7. Have been or are currently suffering from any clinically serious disease of the cardiovascular system, digestive system, respiratory system, endocrine system, nervous system, hematology, immunology, skin, tumor, psychiatric and metabolic abnormalities, or any other disease or physiological condition that can interfere with the test results;
8. The presence of risk factors for Torsade de Pointes (such as a history of heart failure, hypokalemia, or a family history of prolonged QT syndrome), or a history of sick sinus syndrome, or a history of previous myocardial infarction;
9. Patients who have undergone major surgery or whose surgical incision has not fully healed within the 6 months prior to the screening period, including but not limited to any surgery with significant bleeding risk, extended period of general anesthesia or open biopsy or significant traumatic injury (except surgery for recovered appendicitis or proctocele);
10. Severe allergy, including allergy to the investigational drug or any excipient in the investigational drug, allergy to two or more other drugs or food ingredients;
11. Those who have special requirements for diet and cannot comply with a unified diet;
12. Perianal disease with regular/bleeding stool;
13. Habitual constipation or diarrhea, irritable bowel syndrome, inflammatory bowel disease;

    Living habits:
14. Irregular or difficult bowel movements, or other circumstances as assessed by the investigator that affect the collection of stool samples;
15. Binge drinking or regular drinking in the six months preceding the screening period, i.e. drinking more than 14 units of alcohol per week (1 unit =360 mL beer or 45 mL spirits with 40% alcohol or 150 mL wine); Or positive alcohol breath test at screening period;
16. Smokers who smoked more than 5 cigarettes per day or habitually used nicotine-containing products in the 3 months before the screening period and could not quit during the trial;
17. Drug abuse or dependence, urine drug abuse screening positive;
18. Habitual drinking of grapefruit juice or excessive tea (more than 8 cups a day, 1 cup =250 mL), excessive intake of caffeine (more than 3 cups a day coffee, 1 cup =250 mL), and unable to abstain during the trial;

    Others:
19. Workers who require prolonged exposure to radioactive conditions; Or had significant radiation exposure (≥2 chest/abdominal CT, or ≥3 other types of X-rays) within 1 year prior to the test or participated in a radiopharmaceutically labeled test within 1 year;
20. The subject who is fertile has a birth plan or sperm donation plan within 1 year after the signing of the informed consent, or the subject and his or her partner do not agree to take effective contraceptive measures (such as condoms, contraceptive sponges, contraceptive gels, contraceptive membranes, intrauterine devices, oral or injectable contraceptives, subcutaneous implants, etc.);
21. Those who have lost blood or donated blood up to 400 mL within 3 months before the screening period, or received blood transfusions within 1 month;
22. Subjects who have any other factors deemed unsuitable for participation in this study by the investigator.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2024-10-17 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Mean Cumulative Amount of Total Radioactivity (CumAe) of [14C]SIM0270 Excreted in Urine, Feces, and Total (Urine and Feces Combined) Over the Entire Collection Period | From Day 1 to Day 44
  Following a single oral dose of 60 milligrams/150μCi of [14C]SIM0270, urine and fecal samples were collected over time from each participant. The amounts of total radioactivity excreted in the samples were determined using liquid scintillation counting.
Mean Cumulative Amount of Total Radioactivity Expressed as a Percentage of the Radioactive Dose Administered (CumFe) of [14C]SIM0270 Recovered in Urine, Feces, and Total (Urine and Feces Combined) Over the Entire Collection Period | From Day 1 to Day 44
  Following a single oral dose of 60 milligrams/150μCi of [14C]SIM0270, urine and fecal samples were collected over time from each participant. The amounts of total radioactivity excreted in the samples were determined using liquid scintillation counting.
Maximum 0bserved Concentration (Cmax), Estimated for SIM0270 in Plasma and for Total Radioactivity in Plasma | From 0 to 432 hours
  Pharmacokinetic parameters were estimated where possible and appropriate for each participant profile by non-compartmental analysis methods using Phoenix WinNonlin software. Plasma concentrations of SIM0270 were determined using liquid chromatography with tandem mass spectrometry. Total radioactivity concentrations in plasma and whole blood were determined using liquid scintillation counting.
Time to Maximum 0served Concentration (Tmax), Estimated for SIM0270 in Plasma and for Total Radioactivity in Plasma | From 0 to 432 hours
  Pharmacokinetic parameters were estimated where possible and appropriate for each participant profile by non-compartmental analysis methods using Phoenix WinNonlin software. Plasma concentrations of SIM0270 were determined using liquid chromatography with tandem mass spectrometry. Total radioactivity concentrations in plasma and whole blood were determined using liquid scintillation counting.
Area Under the Concentration-Time Curve From Time 0 to 432 Hours AUC(0-432), Estimated for SIM0270 in Plasma and for Total Radioactivity in Plasma | From 0 to 432 hours
  Pharmacokinetic parameters were estimated where possible and appropriate for each participant profile by non-compartmental analysis methods using Phoenix WinNonlin software. Plasma concentrations of SIM0270 were determined using liquid chromatography with tandem mass spectrometry. Total radioactivity concentrations in plasma and whole blood were determined using liquid scintillation counting.
Terminal Elimination Half-Life (t1/2), Estimated for SIM0270 in Plasma and for Total Radioactivity in Plasma | From 0 to 432 hours
  Pharmacokinetic parameters were estimated where possible and appropriate for each participant profile by non-compartmental analysis methods using Phoenix WinNonlin software. Plasma concentrations of SIM0270 were determined using liquid chromatography with tandem mass spectrometry. Total radioactivity concentrations in plasma and whole blood were determined using liquid scintillation counting.

SECONDARY OUTCOMES:
The incidence of Adverse events | From signing ICF until 14 days after departure from the study.
  The incidence and grading of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No